CLINICAL TRIAL: NCT05148728
Title: Prospective Randomized Trial in Low Grade Bladder Tumors: Active Surveillance vs Endoscopic Fulguration.
Brief Title: Active Surveillance vs in Office Fulguration for Low Grade Bladder Cancer Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vall Hebron Insitut Recerca (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR(AG)401/2021
Record Dates: First submitted 2021-11-26; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Bladder Cancer
Keywords: active surveillance; fulguration; bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active surveillance (No Intervention): After a recurrence in patient with previous low grade bladder cancer tumor, strict follow up with cystoscopy and cytology, avoiding immediate surgery
- endoscopic fulguration (Active Comparator): After a recurrence in patient with previous low grade bladder cancer tumor, fulguration under local anesthesia and sedation will be performed using a flexible cystoscope and a monopolar electrode
  Interventions: Procedure: Endoscopic fulguration

INTERVENTIONS:
Procedure: Endoscopic fulguration — already included. WE will use Storz monopolar device for fulguration
  Other Names: Active surveillance
  Arms: endoscopic fulguration

SUMMARY:
Biological behabiour of low grade bladder cancer tumors is well known. They have a very high rate of recurrences during their follow up but very low (less than 1%) risk of progression.

Until now, the gold standard of any bladder recurrence for this patients is performing an immediate transurethral ressection of the tumor.

This surgery has risk of complications and, due to the low risk of these subgroup of tumors, sometimes it becomes an overtreatment for the patients.

This is the reason why new conservative or less invasive surgeries are proposed to follow up and treat these patients.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent Ta-T1a (above muscularis mucosa) LOW GRADE bladder tumor
* Accept cystoscopy surveillance
* Main lession less than 10mm
* Less than 7 lesions
* Negative or low grade cytology
* No solid aspect

Exclusion Criteria:

* previous High grade bladder cancer tumors
* previous Cis
* previous Upper Urinary Tract tumor
* previous pelvic radiotherapy
* hematuria
* meatal localisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Progression rate | two years
  Number of patients that progress during the follow up
Complications rate | two years
  Number and grade of complications in both arms. Clavien Dindo Scale will be used

SECONDARY OUTCOMES:
recurrence rate | two years
  number of recurrences
quality of life measured with CAVICAVENMI questionnaire | two years
  quality of life of the patients in both subgroups. CAVICAVENMI questionnaire will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Fernando Lozano Palacio, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
codified information (anonymous information)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after completing the recruitment (two years), data will be available, for 5 years